CLINICAL TRIAL: NCT03441152
Title: The Neural Effects of Multisession Transcranial Direct Current Stimulation in Older Adults at Risk for Mild Cognitive Impairment and Its Impact in Cognitive Functions and Everyday Memory: A Randomized Controlled Trial
Brief Title: The Effects of Transcranial Direct Current Stimulation in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Kenneth N. K. Fong, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HongKongPUPabloRS
Record Dates: First submitted 2018-02-05; First posted 2018-02-22 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Neuromodulation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS+CT (Experimental): application of tDCS in combination with CT
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): application of sham tDCS in combination with CT
  Interventions: Device: tDCS
- CT (Active Comparator): application of CT
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Transcranial direct current stimulation

SUMMARY:
Objectives: 1) To examine whether the real transcranial direct current stimulation (tDCS) group would perform better in the cognitive training (CT) intervention than the sham tDCS group and the CT group; 2) To determine if, as a consequence of the stimulation generated by the use of tDCS, there would be a transfer effect to other cognitive domains and to cognitive tasks in activities of daily living; 3) To investigate the time and spatial responses of tDCS on the brain cortex during and after tDCS application.

Hypothesis to be tested: By applying anodal tDCS with the combination of a CT delivered via the use of tablet PCs in older adults at risk of MCI, it will enhance their cognitive task performance in CT and subsequently generalize to other cognitive domains as well, involving a transferability to cognitive tasks in activities of daily living.

Design and subjects: A multi-centered single-blinded randomized controlled trial (RCT) with three groups (CT alone/Sham tDCS with the combination of a CT/ Real tDCS coupling with CT) The participants who will take part of this study will be older adults at risk of MCI Study instruments: tDCS, Ipad, Neuron Up CT Apps, EEG. Interventions: The intervention will last for 9 sessions (3 sessions per week for 3 weeks). Sham tDCS and real tDCS, will be combined with the same CT which is used in the CT group. During the experimental intervention, anodal tDCS will be placed on left dorsolateral prefrontal cortex (DLPFC) and cathodal tDCS on the contralateral deltoid muscle with the combination of a CT. During the experimental intervention, anodal tDCS will be placed on left dorsolateral prefrontal cortex (DLPFC) and cathodal tDCS on the contralateral deltoid muscle with the combination of a CT.

Main outcome measures: Cognitive assessments, CT performance, EEG. In addition, delta and theta frequency suppression and alpha increment power under the anode electrode will be observed.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will follow the modified Petersen's criteria:

  1. Aged between 60 and 85 years old;
  2. Obtaining a score on the Montreal Cognitive Assessment Test (MoCA) between 19 and 26;
  3. Achieving a score on the Clinical Dementia Rating (CDR) of 0.5 or below ;
  4. Self-reported cognitive decline by the participants themselves and
  5. Being independent in daily living activities.

     Additional criteria in this study include:
  6. Having completed three or more years of primary education;
  7. Ability to participate in a therapy session lasting at least 30 minutes;
  8. Community ambulant with or without aids; and
  9. Ability to perform a proper range of motion with hands in order to use a tablet PC.

Exclusion Criteria:

* 1) Individuals presenting with a diagnosis of dementia or any other neurological disease; (2) Individuals with depression determined by a score on Geriatric Depression Scale of >5, (3) History of drug or alcohol abuse or dependence in the last 3 months; and (4) Participants who had metallic fixtures around the cephalic area or skin lesions in the areas at where the electrodes were going to be attached were excluded from the study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 10 minutes
  It is a 30-point test about several cognitive domains (visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall and orientation) and a screening tool used of MCI and dementia.
Digit Span Test | 10 minutes
  The test measures short term memory in such a way that sequences of digits are presented and have to be recalled in forward and reverse order. Testing ends when the maximal list length is reached or when subjects fail to recall the trial at one sequence length.
Trial Making Test (TMT) | 5 minutes
  TMT encompasses visual attention and processing speed, it consists of 2 parts in which a set of 25 dots in the first part and 24 dots in the second part have to be accurately connected. Time performance is measured as the main outcome

SECONDARY OUTCOMES:
Riverhead Behavioral Memory Test (3rd edition) (RBMT-3) | 40 minutes
  It includes 14 subtests assessing aspects of visual, verbal, recall, recognition, immediate and delayed everyday memory. Additionally prospective memory skills and the ability to learn new information are measured as well

OTHER OUTCOMES:
Cognitive training activities ( Neuronup cognitive training) | 30 minutes each session ( 9 sessions in total)
  Performance of the cognitive training activities conducted every session
EEG | 15 minutes
  time and spatial responses of tDCS on the brain cortex before and after tDCS application

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gonzalez PC, Fong KNK, Brown T. Transcranial direct current stimulation as an adjunct to cognitive training for older adults with mild cognitive impairment: A randomized controlled trial. Ann Phys Rehabil Med. 2021 Sep;64(5):101536. doi: 10.1016/j.rehab.2021.101536. Epub 2021 Jul 20. PMID 33957292